CLINICAL TRIAL: NCT05308095
Title: Non-randomised, Controlled, Interventional Single-centre Study for the Design and Evaluation of an In-vehicle Hypoglycaemia Warning System in Diabetes The HEADWIND Study Part IV
Brief Title: The HEADWIND Study - Part 4
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Swiss Federal Institute of Technology (Other); University of St.Gallen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HEADWIND 4
Record Dates: First submitted 2022-03-24; First posted 2022-04-01 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
Keywords: Automotive Technology; Hypoglycemia; Hypoglycaemia; Driving; Car
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Hypoglycemia; Carney Complex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental)
  Interventions: Other: Controlled hypoglycaemic state while driving

INTERVENTIONS:
Other: Controlled hypoglycaemic state while driving — Participants will drive on a designated circuit with a real car on a test track accompanied by a driving instructor. Initially, a euglycaemic state (5.0 - 8.0 mmol/L) is established and blood glucose is then declined to hypoglycaemia (3.0 - 3.5 mmol/L) by administering insulin. Thereafter, blood glucose is raised again to euglycaemia (5.0 - 8.0mmol/L). During the procedure, driving data is recorded. Additionally, eye movement, head pose, facial expression, heart rate, skin conductance, and CGM values are recorded throughout the glycemic trajectory. Participants are blinded to the blood glucose values during the procedure.

SUMMARY:
To analyse driving behavior of individuals with type 1 diabetes in eu- and mild hypoglycaemia while driving in a real car. Based on the in-vehicle variables, the investigators aim at establishing algorithms capable of discriminating eu- and hypoglycaemic driving patterns using machine learning classifiers.

DETAILED DESCRIPTION:
Hypoglycaemia is among the most relevant acute complications of diabetes mellitus. During hypoglycaemia physical, psychomotor, executive and cognitive function significantly deteriorate. These are important prerequisites for safe driving.

Accordingly, hypoglycaemia has consistently been shown to be associated with an increased risk of driving accidents and is, therefore, regarded as one of the relevant factors in traffic safety. Therefore, this study aims at evaluating a machine-learning based approach using in-vehicle data to detect hypoglycaemia during driving.

During controlled eu- and hypoglycaemia, participants with type 1 diabetes mellitus drive in a driving school car on a closed test-track while in-vehicle data is recorded. Based on this data, the investigators aim at building machine learning classifiers to detect hypoglycemia during driving.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent as documented by signature
* Type 1 Diabetes mellitus as defined by WHO for at least 1 year or confirmed C-peptide negative (<100pmol/l with concomitant blood glucose >4 mmol/l)
* Age between 21-60 years
* HbA1c ≤ 9.0 %
* Functional insulin treatment with good knowledge of insulin self-management
* Passed driver's examination at least 3 years before study inclusion. Possession of a valid, definitive Swiss driver's license.
* Active driving in the last 6 months.

Exclusion Criteria:

* Contraindications to the drug used to induce hypoglycaemia (insulin aspart), known hypersensitivity or allergy to the adhesive patch used to attach the glucose sensor.
* Pregnancy or intention to become pregnant during the course of the study, lactating women or lack of safe contraception
* Other clinically significant concomitant disease states as judged by the investigator
* Physical or psychological disease likely to interfere with the normal conduct of the study and interpretation of the study results as judged by the investigator
* Renal failure
* Hepatic dysfunction
* Coronary heart disease
* Other cardiovascular disease
* Epilepsy
* Drug or alcohol abuse
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant
* Participation in another study with an investigational drug within the 30 days preceding and during the present study
* Total daily insulin dose >2 IU/kg/day
* Specific concomitant therapy washout requirements prior to and/or during study participation
* Current treatment with drugs known to interfere with metabolism or driving performance

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2022-04-13 (Actual); Primary Completion 2022-06-23 (Actual); Study Completion 2022-06-23 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of the hypoglycaemia warning system using in-vehicle data to detect hypoglycaemia quantified as the area under the receiver operating characteristics curve (AUROC). | 240 minutes
  The machine learning model is developed and evaluated based on in-vehicle data generated in eu- and hypoglycaemia. Detection performance of hypoglycaemia is quantified as AUROC.

SECONDARY OUTCOMES:
Diagnostic accuracy of the hypoglycaemia warning system using wearable data to detect hypoglycaemia quantified as the area under the receiver operating characteristics curve (AUROC). | 240 minutes
  The machine learning model is developed and evaluated based on wearable data recorded in eu- and hypoglycaemia. Detection performance of hypoglycemia is quantified as AUROC.
Diagnostic accuracy of the hypoglycaemia warning system using in-vehicle data and recordings of the continous glucose monitoring (CGM) system to detect hypoglycaemia quantified as sensitivity and specificity. | 240 minutes
  The CGM device is in use during controlled eu- and hypoglycaemia. Detection performance of hypoglycaemia is quantified as sensitivity and specificity.
Diagnostic accuracy of the hypoglycaemia warning system using wearable data and recordings of the CGM system to detect hypoglycaemia quantified as sensitivity and specificity. | 240 minutes
  The CGM device is in use during controlled eu- and hypoglycaemia. Detection performance of hypoglycaemia is quantified as sensitivity and specificity.
Change in driving features over the glycaemic trajectory. | 240 minutes
  Driving signals are recorded using a driving simulator.
Change of gaze coordinates over the glycaemic trajectory. | 240 minutes
  Gaze coordinates are recorded using an eye-tracker device.
Change of head pose over the glycaemic trajectory. | 240 minutes
  Head pose (position/rotation) is recorded using an eye-tracker device.
Change of heart rate over the glycaemic trajectory | 240 minutes
  Heart rate is recorded using a holter-ECG device and a wearable.
Change of heart rate variability over the glycaemic trajectory | 240 minutes
  Heart rate variability is recorded using a holter-ECG device and a wearable.
Change of electrodermal activity over the glycaemic trajectory | 240 minutes
  Electrodermal activity is recorded using a wearable.
Hypoglycaemic symptoms over the glycaemic trajectory. | 240 minutes
  Hypoglycemic symptoms are rated using a validated questionnaire (minimum score = 0, maximum score = 6, a higher score means more symptoms)
Change of cognitive performance over the glycaemic trajectory. | 240 minutes
  Cognitive performance will be assessed using the Trail Making B Test (lower time in seconds means better performance) and using the Digital Symbol Substitution Test (higher score means better performance).
Time course of the hormonal response over the glycaemic trajectory | 240 minutes
  Epinephrine, norepinephrine, glucagon, cortisol and growth hormone will be measured at pre-defined time points.
Self assessment of driving performance over the glycaemic trajectory. | 240 minutes
  Participants rate their driving performance on a 7-point Likert Scale (lower value means poorer driving performance).
Number of driving mishaps over the glycaemic trajectory. | 240 minutes
  Any driving mishaps, accidents and interventions by the driving instructor will be documented.
CGM accuracy over the glycaemic trajectory | 240 minutes
  CGM values will be recorded using a CGM sensor. Venous blood glucose is considered as the reference. Accuracy will be quantified using mean absolute relative difference (MARD) from the gold-standard and using the Clarke error grid.
Accuracy of our protocol to induce hypoglycaemia in achieving the intended hypoglycaemic range. | 240 minutes
  Accuracy will be quantified using mean absolute relative difference from the intended hypoglycaemic range.
Number of Adverse Events (AEs) | 2 weeks, from screening to close out visit in each participant
  Adverse Events will be recorded at each study visit.
Number of Serious Adverse Events (SAEs) | 2 weeks, from screening to close out visit in each participant
  Serious Adverse Events will be recorded at each study visit.
Emotional response to the hypoglycaemia warning system | 240 minutes
  Physiological response will be measured using an electro-dermal activity sensor (skin conductance) and eye tracker (eye blinks). Self-reported emotional response will be assessed with scales (e.g., valence, arousal, annoyance, sense of urgency).
Technology acceptance of the hypoglycaemia warning system | 240 minutes
  Technology acceptance will be measures with user experience questionnaires, such as the Unified Technology Acceptance and Use of Technology Questionnaire and free words associations.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Stettler, Prof. MD, Principal Investigator — Inselspital, Bern University Hospital, University of Bern, Switzerland, Department of Diabetes, Endocrinology, Nutritional Medicine and Metabolism, Bern, Switzerland
Locations (1):
- University Department of Endocrinology, Diabetology, Clinical Nutrition and Metabolism, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Any requests for raw data will be reviewed by the HEADWIND scientific study board comprising the principal investigator (PI) and Co-PI as well as senior researchers leading the involved research groups at University Hospital Bern, Swiss Federal Institute of Technology (ETH) Zurich, and University of St. Gallen. Only applications for non-commercial use will be considered and should be sent to the PI. Applications should outline the purpose for the raw-data transfer. Any data that can be shared will need approval from the HEADWIND scientific study board and a Material Transfer Agreement in place. All data shared will be de-identified.
Supporting Information: Analytic Code
Access Criteria: Only applications for non-commercial use will be considered and should be sent to the PI.

REFERENCES:
- [Derived] Berube C, Maritsch M, Lehmann VF, Kraus M, Feuerriegel S, Zuger T, Wortmann F, Stettler C, Fleisch E, Kocaballi AB, Kowatsch T. Multimodal In-Vehicle Hypoglycemia Warning for Drivers With Type 1 Diabetes: Design and Evaluation in Simulated and Real-World Driving. JMIR Hum Factors. 2024 Apr 18;11:e46967. doi: 10.2196/46967. PMID 38635313